CLINICAL TRIAL: NCT06293547
Title: Clinical Effectiveness and Parental Acceptance of Silver Diamine Fluoride in Preschool Children: A Non-randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, BURAK BULDUR, Professor of Pediatric Dentistry, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIS-2022-295
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Silver Diamine Fluoride
Keywords: caries, silver daimine fluoride, primary teeth
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: The study group of this non-randomized, prospective, single-arm clinical research consisted of pediatric patients and their parents who presented to the Department of Pediatric Dentistry, Faculty of Dentistry, Cumhuriyet University, selected using convenient sampling method. For determining the sample size in this study, assuming a 5% alpha error, 80% power, and a cessation rate (35.7%) from a previous study, it was calculated that at least 40 participants should be included. Considering potential patient loss/follow-up, the study group was increased by 20%, resulting in a final decision to include 48 children and their parents in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Following a standard dental examination, which may have included intraoral radiographs as needed, the application of 38% SDF (Riva Star, SDI Australia) was conducted on carious lesions identified in primary teeth. The application procedure of SDF adhered to the protocol recommended in the literature and the instructions provided by the manufacturer. One and experienced researcher applied SDF to each patient. Initially, the affected teeth were isolated and dried using gauze and cotton rolls. Subsequently, the SDF solution was applied directly to the lesions using a microbrush, with an absorption time ranging from a minimum of 30 seconds to a maximum of 120 seconds, depending on the child's behavior (30-60-90-120 seconds). Any excess solution was carefully removed using gauze. Parents were instructed to ensure that the child refrained from eating or drinking for at least one hour following the application of SDF.
  Interventions: Drug: Silver Diamine Fluoride

INTERVENTIONS:
Drug: Silver Diamine Fluoride — Silber Diamine Fluoride, a colorless, odorless alkaline solution, effectively halts carious lesions in various populations, including children and elderly patients, or those averse to invasive treatments. Its high fluoride content facilitates remineralization, caries arrest, and prevention. SDF application is simple, non-invasive, cost-effective, and does not stain intact enamel, making it suitable for treating dentin hypersensitivity. Its ease of use is advantageous for children, patients with special needs, and the elderly. Particularly beneficial for high-risk patients with salivary dysfunction or multiple carious lesions, SDF offers potential in pediatric dentistry and community oral health by streamlining procedures, requiring rapid application without sharp instruments or anesthesia.
  Other Names: SDF

SUMMARY:
Silver diamine fluoride (SDF) is a topical fluoride agent that has emerged in recent years and has a strong potential to arrest dentinal caries in early childhood caries. SDF has been developed as an effective non-invasive treatment method, especially in the non-cooperative preschool group, with its advantages such as easy application, low cost, and limited technical difficulties. The aims of this study were as follow: (a) to evaluate the efficacy of 38% GDF in arresting active dental caries lesions and reducing or preventing associated dental pain and infections in at-risk young children; and (b) how SDF treatment is perceived and acceptable by parents. The null hypothesis of the study was that 38% SDF treatment will be effective in arresting active dental caries lesions and reducing the incidence of pain and infection in young children, and is well-accepted by parents. The study group of this clinical research will consist of pediatric patients and their parents who were selected by easily accessible case sampling method and applied to Sivas Cumhuriyet University Faculty of Dentistry Pediatric Dentistry clinic. The working group will consist of a total of 48 children and their parents who meet the inclusion criteria. Parents will also be briefed on the GDF, follow-up instructions, oral hygiene instructions, and dietary education. After a baseline examination including radiographs taken during a standard dental examination, 38% GDF will be applied to carious lesions detected in primary teeth. Carious lesions will be treated with 38% SDF application once or twice. Children will be reassessed at 3-week, 3-month and 6-month follow-up sessions to assess color and structural changes in carious lesions (soft/hard). Parents will be asked to answer a questionnaire including questions about pain or infection symptoms and their views on SDF treatment.

DETAILED DESCRIPTION:
Ethical Approval Clinical examination and data collection procedures were conducted at the Department of Pediatric Dentistry, Faculty of Dentistry, Cumhuriyet University, following ethical approval from the Clinical Research and Ethics Committee of Sivas Cumhuriyet University Medical Faculty on June 14, 2022 (Approval No: 2022-06/04). All parents or legal guardians of the children participating in the study were provided with information about the study prior to the procedures, and signed informed consent forms were obtained.

Research Design The study group of this non-randomized, prospective, single-arm clinical research consisted of pediatric patients and their parents who presented to the Department of Pediatric Dentistry, Faculty of Dentistry, Cumhuriyet University, selected using convenient sampling method. For determining the sample size in this study, assuming a 5% alpha error, 80% power, and a cessation rate (35.7%) from a previous study, it was calculated that at least 40 participants should be included. Considering potential patient loss/follow-up, the study group was increased by 20%, resulting in a final decision to include 48 children and their parents in the study. The CONSORT (Consolidated Standards of Reporting Trials) flow diagram showing the research design and protocol is depicted in Figure 1.

Inclusion and Exclusion Criteria The inclusion criteria for the study were as follows: voluntary participation, mentally and physically healthy children aged 3-5 years, and mentally and physically healthy parents with native literacy. Children having at least one carious lesion identified according to International Caries Detection and Assessment System (ICDAS) criteria to be included in the study. Lesions classified using the ICDAS scale are as follows: active (soft) cavitated carious lesions extending into dentine during primary dentition (ICDAS 5 or 6); non-cavitated lesions (ICDAS 3 or 4); or initial carious lesions (ICDAS 1 or 2). Those with ICDAS scores of 3, 4, 5, and 6 were included in the study. The exclusion criteria for the current study were as follows: small interproximal caries not clinically observable; children showing signs of spontaneous pain, tooth mobility, or pulp infection due to caries; medical issues preventing treatment in the clinic, congenital developmental defects, allergies or sensitivities to SDF, and non-cooperation or failure to attend follow-up visits.

SDF Applicaiton Informed consent was obtained from the parents or legal guardians of the children participating in the study. Additionally, detailed information SDF treatment, follow-up instructions, oral hygiene guidelines, and dietary education was provided to the parents. Following a standard dental examination, which may have included intraoral radiographs as needed, the application of 38% SDF (Riva Star, SDI Australia) was conducted on carious lesions identified in primary teeth. The application procedure of SDF adhered to the protocol recommended in the literature and the instructions provided by the manufacturer. One and experienced researcher applied SDF to each patient. Initially, the affected teeth were isolated and dried using gauze and cotton rolls. Subsequently, the SDF solution was applied directly to the lesions using a microbrush, with an absorption time ranging from a minimum of 30 seconds to a maximum of 120 seconds, depending on the child's behavior (30-60-90-120 seconds). Any excess solution was carefully removed using gauze. Parents were instructed to ensure that the child refrained from eating or drinking for at least one hour following the application of SDF.

The isolation of the lesion is vital component of the protocol, ensuring the efficacy of SDF in arresting the progression of the lesion. Therefore, children were scheduled for follow-up appointments at 3 weeks, 3 months and 6 months (recall visits) to assess the status of the lesions. If the carious lesions did not exhibit characteristics of being black and hard at both recall appointments, indicating non-progression, a second application of SDF was administered.

Documentation of the SDF treatment applied at each appointment was meticulously maintained. The study concluded either upon the completion of treatment in the clinic or when active carious lesions were effectively arrested, and the child's cooperation and behavior improved during follow-up visits. Subsequent to confirming the cessation of carious lesions at the final treatment stage, appropriate restorative procedures were planned for both anterior and posterior teeth, as indicated.

Patients who exhibited difficulty in cooperation were either scheduled for routine follow-up visits or referred for treatment under sedation or general anesthesia, depending on the severity of the case and the patient's needs.

Data Collection Primary Outcome The primary outcome was evaluating the efficacy of SDF treatment in arresting active carious lesions. This assessment was conducted through clinical examinations of the patients.

Clinical Assessment of Arrested Caries Lesions A standardized control form was utilized for clinical evaluation. Treatment and follow-up procedures were conducted by a single experienced and trained pediatric dentist (BB). The color of dentin (yellow, black, brown) and the texture of lesions (soft, hard, chalky, shiny) were assessed and noted using a dental probe with light pressure at the initial visit and at each follow-up session. The presence or absence of pain and infection was recorded at baseline and during each follow-up session using clinical examination and parental interviews. The effectiveness of SDF was assessed through clinical outcomes, with dark, hard, and black lesions without pain or infection considered positive outcomes. Signs indicating treatment failure included lesion progression, a yellow, soft lesion, or the presence of pain or infection.

The total application time for each SDF treatment was documented in seconds. The duration was set between a minimum of 30 seconds and a maximum of 120 seconds for each tooth.

Secondary Outcome The secondary outcome was to assess parental acceptance of SDF treatment. This evaluation was carried out using a questionnaire that had been validated previously.

Parental Perceptions of Silver Diamine Fluoride Dental Color Changes Questionnaire The acceptability of SDF treatment by parents was measured using the Parental Perceptions of Silver Diamine Fluoride Dental Color Changes Questionnaire filled out by parents before treatment and at the 6-month follow-up appointments. The Silver Diamine Fluoride Dental Color Change Parent Perception Survey, developed by Crystal et al., has an original English version. The survey utilizes a closed-ended Likert scale type of questions, presenting a series of full-color photographs showing anterior and posterior primary teeth before and after SDF treatment to gather parental opinions based on visual observation. The Turkish validation of the scale has been previously conducted.

The survey is distributed into 3 subscales comprising a total of 14 items: (a) overall acceptability based on staining effects only on posterior (item 1) and anterior (item 2) teeth; acceptability in a positive child cooperation scenario (items 3-4: cooperative child; items 5-6: child upset but cooperative); and acceptability in a negative child cooperation scenario with increased barriers to traditional restorations (items 7-8: child crying; items 9-10: child screaming or kicking; items 11-12: need for oral sedation; and items 13-14: need for general anesthesia). Parents are asked to provide separate responses for anterior and posterior teeth for each scenario. Response options and scoring for items 1-2 are as follows: "unacceptable" (1 point); "partially unacceptable" (2 points); "partially acceptable" (3 points); and "acceptable" (4 points). For items 3-14, response options and scoring are as follows: "definitely not possible" (score 1); "not very possible" (score 2); "partially possible" (score 3); and "very possible" (score 4). Specific scores for domains are calculated by averaging the scores of the items within each domain for both anterior and posterior teeth. Higher average scores indicate higher acceptability for SDF staining.

The acceptability of SDF treatment by parents was measured by completing the relevant survey face-to-face before treatment and at the 6-month follow-up appointment.

Socio-demographic and oral health behaviors form Parents were provided with a socio-demographic and oral health behaviors survey form aimed at measuring socioeconomic status and oral health behaviors. The validation of the form had been previously conducted. The form included questions regarding parental educational level, income status, health insurance, frequency of tooth brushing, frequency of dental visits, the last time they visited a dentist, and negative dental experiences. Additionally, parents were asked about their children's gender, age, time and frequency of consuming cariogenic foods, frequency of tooth brushing, frequency of dental visits, the last time their child visited a dentist, and negative dental expreinces.

Statistical Analysis The data were analysed using SPSS software (Ver.24, IBM Corp., Armonk, NY). Descriptive statistics (frequency and percentage, or mean and standard deviation) were used to describe the demographic characteristics and socioeconomic status of both children and parents.

The chi-square test was employed to assess the relationship between the durations of SDF applications and the cessation of lesion progression. To evaluate the effectiveness of arresting lesion progression, the proportion of lesions that did not progress before and after SDF application was calculated. Fisher's exact chi-square test was used for categorical variables.

Continuous variables were tested for normal distribution using the Shapiro-Wilk test. Repeated measures analysis of variance (ANOVA) was conducted to examine the effects of treatment and various variables related to children and parents' sociodemographic and oral health behaviors. Paired samples t-test was utilized for comparing pre-test and post-test values within groups. A P-value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the study were as follows: voluntary participation, mentally and physically healthy children aged 3-5 years, and mentally and physically healthy parents with native literacy. Children having at least one carious lesion identified according to International Caries Detection and Assessment System (ICDAS) criteria to be included in the study. Lesions classified using the ICDAS scale are as follows: active (soft) cavitated carious lesions extending into dentine during primary dentition (ICDAS 5 or 6); non-cavitated lesions (ICDAS 3 or 4); or initial carious lesions (ICDAS 1 or 2). Those with ICDAS scores of 3, 4, 5, and 6 were included in the study.

Exclusion Criteria:

The exclusion criteria for the current study were as follows: small interproximal caries not clinically observable; children showing signs of spontaneous pain, tooth mobility, or pulp infection due to caries; medical issues preventing treatment in the clinic, congenital developmental defects, allergies or sensitivities to SDF, and non-cooperation or failure to attend follow-up visits.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical Assessment of Arrested Caries Lesions | 6 month
  The primary outcome was evaluating the efficacy of SDF treatment in arresting active carious lesions. This assessment was conducted through clinical examinations of the patients.

SECONDARY OUTCOMES:
Parental acceptance of SDF treatment | 6 month
  The acceptability of SDF treatment by parents was measured using the Parental Perceptions of Silver Diamine Fluoride Dental Color Changes Questionnaire filled out by parents before treatment and at the 6-month follow-up appointments. The Silver Diamine Fluoride Dental Color Change Parent Perception Survey, developed by Crystal et al., has an original English version. The survey utilizes a closed-ended Likert scale type of questions, presenting a series of full-color photographs showing anterior and posterior primary teeth before and after SDF treatment to gather parental opinions based on visual observation

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No